CLINICAL TRIAL: NCT03080259
Title: Primary Care Prevention of Stimulant Diversion by High School Students With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Brooke S. G. Molina, Ph.D., Professor of Psychiatry and Psychology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U01DA040213 (NIH); U01DA040213 (NIH)
Record Dates: First submitted 2016-06-17; First posted 2017-03-15 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: ADHD
Keywords: ADHD; Stimulant Misuse; Stimulant Diversion
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulant Diversion Prevention (Active Comparator): Providers will be trained in methods to prevent or decrease the likelihood of stimulant diversion by their adolescent patients (education and counseling, strategies for use by patients and parents, and treatment adjustments).
  Interventions: Behavioral: Stimulant Diversion Prevention (SDP)
- Treatment As Usual (No Intervention): Standard clinical care

INTERVENTIONS:
Behavioral: Stimulant Diversion Prevention (SDP) — provider training, patient/parent education and counseling, strategies for use by patients and parents, and treatment adjustments
  Arms: Stimulant Diversion Prevention

SUMMARY:
The purpose of this study is to test clinical strategies that pediatric providers may use to prevent misuse and diversion of stimulants by their adolescent patients with ADHD.

DETAILED DESCRIPTION:
This study addresses the increase in diversion (selling, sharing, loaning, or trading) of prescription stimulant medications by adolescents with Attention-Deficit/Hyperactivity Disorder (ADHD). In the absence of any standardized, empirically evaluated clinical strategies or interventions to prevent or decrease stimulant diversion, this project will test the effect of a brief provider-led intervention for stimulant diversion prevention among adolescents being prescribed stimulant medication in pediatric care. The investigators hypothesize that adolescents treated in pediatric practices randomized to the intervention will report decreased diversion, increased perceived risk of harm, and decreased intentions to divert compared to adolescents treated in pediatric practices randomized to treatment-as-usual. Secondary analyses will examine the effect of the intervention on additional contributing variables (e.g., patient, parent, and provider attitude and behavior change).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD
* Treatment with stimulant medication
* Enrolled in or attending middle school or high school
* Parent/guardian willing to participate
* Receiving treatment at one of the 7 pediatric practices participating in the protocol

Exclusion Criteria:

* Not diagnosed with ADHD
* Not treated with stimulant medication
* Not enrolled or attending middle school or high school
* Parent/guardian unwilling to participate
* Not receiving treatment at one of the 7 pediatric practices participating in the protocol

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 357 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Diversion Activity Questionnaire (Diversion); Change from baseline across follow-up assessments | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Items indicating frequency (# of times) selling, sharing, trading, or loaning stimulant medication. Diversion frequency will increase less in the SDP group between baseline and follow-up assessments.
Perceived Risk of Harm Questionnaire; Change from baseline across follow-up assessments | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Items measuring the degree to which participants believe that people risk harming themselves if they take ADHD medication without a prescription (responses range from "no risk" to "great risk"). Mean perceived harm will increase more after baseline for the SDP vs control group.
Intentions to Divert Prescription Stimulants Questionnaire; Change from baseline across follow-up assessments | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Items measuring intention to share/sell/trade stimulant medication (responses range from "I definitely will" to "I definitely will not"). Intent to divert will increase less in the SDP vs control group.

SECONDARY OUTCOMES:
Utilization of Clinical Practice Strategies for Diversion Prevention Questionnaire | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Items measuring teen's report of the frequency of provider utilization of stimulant diversion prevention techniques (responses range from "no" to "yes, more than once" in the last 6 months). Number of techniques endorsed as occurring at least once will increase. Number will increase after baseline more for the SDP than control group.
Disclosure of Stimulant Treatment Questionnaire | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Number of people and/or groups who know about the teen's ADHD medication prescription (sum total across items). Total number will decrease after baseline in the SDP vs control group.
Diversion Activity Questionnaire (Approaches) | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Number of times approached to sell or share ADHD prescription medication. Number will decrease after baseline more for the SDP than control group.
Management of Peer Requests Questionnaire (Diversion Refusal Skills) | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Increased likelihood (from "definitely not" to "definitely") of using diversion refusal skills. Score will increase after baseline more for the SDP than control group.
Management of Peer Requests Questionnaire (Diversion Refusal Self Efficacy) | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Increased ease (from "very difficult" to "very easy") in perceived use of diversion refusal skills. Score will increase after baseline more for the SDP than control group.
Management of Peer Requests Questionnaire (Diversion Refusal Frequency) | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Increased frequency (from "never" to "almost always") of using diversion refusal skills. Frequency will increase more after baseline for the SDP vs control group.
Knowledge of Stimulant Diversion Consequences Questionnaire | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Items measuring knowledge of negative consequences of diversion; mean score will increase (responses for each consequence ranges from "very unlikely" to "likely"). Mean score will increase after baseline more for the SDP than control group.
Likelihood of Diversion Scale | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Assesses likelihood (response scale ranges from "I definitely would" to "I definitely would not") of diverting medication in specific situations. Mean response across items should increase toward "I definitely would not". Likelihood of diversion mean score will change after baseline toward "I definitely would not" more for the SDP than control group.
Approval of Diversion by Proximal Social Contacts Questionnaire | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Items measuring approval of diversion by proximal social contacts; responses range from "strongly approve" to "strongly disapprove". Mean score will increase towards disapproval. Mean score will increase toward disapproval more for the SDP than control group.
Parental Supervision and Monitoring Specific to ADHD Medication Questionnaire (Attempted) | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Items measuring attempted parental monitoring of stimulant medication (e.g., During the last 6 months, how much did either of your parents try to know.......). Mean score of responses across items. Mean score will increase after baseline more for the SDP than control group.
Parental Supervision and Monitoring Specific to ADHD Medication Questionnaire (Actual) | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Items measuring actual parental knowledge of teen's stimulant medication (e.g., During the last 6 months, how much did either of your parents really know.......). Mean score of responses across items. Mean score will increase after baseline more for the SDP than control group.
Parent-Teen Communication about Alcohol, Drugs, Diversion | baseline, 6 month follow-up, 12 month follow-up, 18 month follow-up
  Items assessing frequency of parent-teen discussion about diversion-related behavior (e.g., "Within the last 6 months, my parents talked with me about keeping my ADHD diagnosis and ADHD medication private"). Responses range from "never" to "three or more times". Number of items endorsed as occurring at least once or more often will increase after baseline more for the SDP than control group.

CONTACTS AND LOCATIONS:
Overall Officials: Brooke SG Molina, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Youth and Family Research Program, WPIC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make de-identified data available to potential scientific collaborators upon request as allowed by local Institutional Review Board (IRB) regulations and after the main findings of the study have been accepted for publication. The investigators will honor requests to use data for research or teaching purposes only and that include a commitment to protect the privacy and confidentiality of the data per IRB requirements. Depending upon the size of the request, the investigators will charge, as needed, reasonable costs associated with preparation of datasets and assistance with dataset utilization.

REFERENCES:
- [Result] Molina BSG, Joseph HM, Kipp HL, Lindstrom RA, Pedersen SL, Kolko DJ, Bauer DJ, Subramaniam GA. Adolescents Treated for Attention-Deficit/Hyperactivity Disorder in Pediatric Primary Care: Characterizing Risk for Stimulant Diversion. J Dev Behav Pediatr. 2021 Sep 1;42(7):540-552. doi: 10.1097/DBP.0000000000000923. PMID 33908377
- [Result] McGuier EA, Kolko DJ, Joseph HM, Kipp HL, Lindstrom RA, Pedersen SL, Subramaniam GA, Molina BSG. Use of Stimulant Diversion Prevention Strategies in Pediatric Primary Care and Associations With Provider Characteristics. J Adolesc Health. 2021 Apr;68(4):808-815. doi: 10.1016/j.jadohealth.2020.12.006. Epub 2021 Jan 11. PMID 33446402
- [Derived] McGuier EA, Kolko DJ, Pedersen SL, Kipp HL, Joseph HM, Lindstrom RA, Bauer DJ, Subramaniam GA, Molina BSG. Effects of Training on Use of Stimulant Diversion Prevention Strategies by Pediatric Primary Care Providers: Results from a Cluster-Randomized Trial. Prev Sci. 2022 Oct;23(7):1299-1307. doi: 10.1007/s11121-022-01411-2. Epub 2022 Aug 11. PMID 35951253